CLINICAL TRIAL: NCT05056506
Title: A Comparison of Limited Endoscopic Sphincterotomy With Endoscopic Papillary Large Balloon Dilation vs. Endoscopic Papillary Large Balloon Dilation for Endoscopic Choledocholithiasis
Brief Title: EPLBD With Limited EST vs. EPLBD for Choledocholithiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jianfeng Yang (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); The Second Affiliated Hospital of Jiaxing University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Shanghai Fourth People's Hospital Tongji University (Other)
Responsible Party: Sponsor-Investigator, Jianfeng Yang, Professor, First People's Hospital of Hangzhou
Organization: First People's Hospital of Hangzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-02-01
Record Dates: First submitted 2021-09-20; First posted 2021-09-24 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Choledocholithiasis
Keywords: Endoscopic sphincterotomy; Endoscopic papillary balloon dilation; Complication; Safety; Choledocholithiasis
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic papillary large balloon dilation group (Active Comparator): Endoscopic papillary large balloon dilation to extract bile duct stones
  Interventions: Procedure: EPLBD
- Endoscopic papillary Large balloon dilation combined with limited endoscopic sphincterotomy group (Experimental): Endoscopic papillary large balloon dilation combined with limited endoscopic sphincterotomy to extract bile duct stones
  Interventions: Procedure: ELPBD+ESD

INTERVENTIONS:
Procedure: EPLBD — Endoscopic papillary large balloon dilation for Choledocholithiasis
  Arms: Endoscopic papillary large balloon dilation group
Procedure: ELPBD+ESD — Endoscopic papillary balloon dilation combined with limited endoscopic sphincterotomy for Choledocholithiasis
  Arms: Endoscopic papillary Large balloon dilation combined with limited endoscopic sphincterotomy group

SUMMARY:
Endoscopic papillary balloon dilation (EPBD) for choledocholithiasis is known to be comparable to endoscopic sphincterotomy (EST) especially in cases of small stones. With larger stones (> 10 mm), EPBD with conventional balloon, which have a diameter of 6-8 mm, was reported as less effective for extraction of stones, requiring additional mechanical lithotripsy (ML). The present study aims to compare the efficacy and safety of limited EST plus endoscopic papillary balloon dilation (EST-EPBD) with endoscopic papillary large balloon dilation for large choledocholithiasis.

DETAILED DESCRIPTION:
ERCP is the best option to remove bile duct stones. It can be done by either endoscopic sphincterotomy (EST) or endoscopic papillary balloon dilation (EPBD). Large bile duct stones appear to be more difficult to remove with conventional methods, such as EST and EPBD. Therefore, extraction of large bile duct stones may require mechanical lithotripsy (ML) as an adjunctive procedure. The primary complication of ML is basket and stone impaction, which can lead to complications such as pancreatitis and cholangitis. Some recent studies have reported the efficacy of endoscopic papillary large balloon dilation (EPLBD) alone or combined with limited EST, establishing it as a safe treatment for the removal of large bile duct stones. The investigators conducted the present study to compare the therapeutic outcome and complications between EPLBD alone and limited EST plus EPLBD for the treatment of large bile duct stones.

ELIGIBILITY:
Inclusion Criteria:

* large bile duct stones (≥10 mm)

Exclusion Criteria:

* pregnancy
* refusal of written informed consent
* Patients with benign or malignant biliary stricture
* Contraindications to ERCP exist
* Complicated with acute pancreatitis or acute cholangitis
* Coagulation dysfunction，thrombocytopenia
* prior EST or EPBD
* Patients after gastrointestinal reconstruction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of complications | within 1 months after the procedure
  The incidence of complications

SECONDARY OUTCOMES:
The success rate of 1st session treatment | within 1 months after the procedure
  The success rate of 1st session treatment
The rate of mechanical lithotripsy | within 1 months after the procedure
  The rate of mechanical lithotripsy
Total ercp times | within 1 months after the procedure
  Total ercp numbers
Overall successful stone removal rate | within 1 months after the procedure
  Overall successful stone removal rate

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, Principal Investigator — Zhejiang University
Locations (2):
- China (2):
  - Shanghai Fourth People's Hospital, Shanghai, Shanghai Municipality
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hwang JC, Kim JH, Lim SG, Kim SS, Shin SJ, Lee KM, Yoo BM. Endoscopic large-balloon dilation alone versus endoscopic sphincterotomy plus large-balloon dilation for the treatment of large bile duct stones. BMC Gastroenterol. 2013 Jan 17;13:15. doi: 10.1186/1471-230X-13-15. PMID 23324454